CLINICAL TRIAL: NCT00263900
Title: Exploratory Study of the Use of the Quick Diagnostic Test of the Influenza and the Infection With RSV by the Paediatric Emergency Unit and Their Impact on the Assumption of Responsibility of the Suspect Children of a Viral Infection
Brief Title: TGV:Use of the Quick Diagnostic Test of the Influenza and the Infection With RSV by the Paediatric Emergency Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Mr François TEILLARD, Research and Innovation Director, Direction de la Recherche et de l'Innovation
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/078/HP
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Influenza; Respiratory Syncytial Viruses
Keywords: Influenza A; Influenza B; RSV
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RSV respi-strip and Quick-vue influenza — Assessments of 2 quick diagnostic tests in the emergency unit during children's care

SUMMARY:
The aim of this study is to evaluate the impact of the use of a quick diagnostic test of infection with RSV and influenza virus on the assumption of clinical responsibility of the children consulting at the Paediatric Emergency Unit.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 5 years
* Isolated fever and/or
* Infection of the higher air routes (congestive otitis, feverish rhinitides, tracheitis or laryngitis) and/or infection of the lower air routes (cough, pneumonia, bronchitis, asthma)
* Signed consent form

Exclusion Criteria:

* Evocative clinical of a urinary and/or bacterial infection
* Purulent acute otitis media
* Typical acute bronchiolitis
* Suspicion of acute lobar pneumonia
* Acute gastro-enteritis
* Anginas
* Serious chronic respiratory pathology
* Other infection whose etiologic viral diagnosis is established
* Congenital or acquired immunizing deficits
* Congenital cardiopathy

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assessments of quick diagnostic test of the Influenza virus and the SRV to measure the utility and the impact of those tests on the care of children in emergency unit | time of support at the emergnecy unit

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARGUET, Professor, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Urgences pédiatriques, Amiens
  - Urgences pédiatriques CHU de Caen, Caen
  - POSU pediatrique, Le Havre
  - Urgences pédiatriques - CHU ROUEN, Rouen